CLINICAL TRIAL: NCT01551628
Title: A Pilot Study of the Safety and Preliminary Efficacy of Recombinant Human Arginase 1 (rhArg1) in Patients With Relapsed or Refractory Leukemia or Lymphoma
Brief Title: A Pilot Study of Recombinant Human Arginase 1 (rhArg1) in Patients With Relapsed or Refractory Leukemia or Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow patient recruitment
Sponsor: Bio-Cancer Treatment International Limited (Industry)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCT-100-003
Record Dates: First submitted 2012-02-29; First posted 2012-03-13 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2014-03

CONDITIONS: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — BCT-100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombinant Human Arginase 1 Peg5000 (Experimental)
  Interventions: Drug: Recombinant human arginase 1 Peg5000

INTERVENTIONS:
Drug: Recombinant human arginase 1 Peg5000 — Patients will receive weekly IV infusions of PEG-BCT-100, until evidence of disease progression, intolerable adverse events, or withdrawal of patient consent. For safety sake, each subject will receive an induction dose of PEG-BCT-100 500 U/kg and 1000 U/kg at week -2 and week -1, respectively. The study dose of PEG-BCT-100 1600 U/kg will be initiated at week 1 (Day1). Each escalation of dose level will be determined by the investigator according to each subject's tolerability and criteria for treatment discontinuation.
  Other Names: PEG-BCT-100, rhArg1peg5000

SUMMARY:
The purpose of this study is to determine whether Recombinant Human Arginase 1 (rhArg1)is safe and effective in the treatment of patients with Relapsed or Refractory Leukemia or Lymphoma.

DETAILED DESCRIPTION:
This is a pilot, open-label study of PEG-BCT-100 in patients with relapsed/refractory leukemia or lymphoma who have satisfied all inclusion/exclusion criteria.

Approximately 15 subjects will be enrolled or when 10 evaluable subjects are included in the study. Evaluable subjects are defined as subjects who have received 4 consecutive doses of PEG-BCT-100 1600U/kg within 6 weeks from the first 1600U/kg dose and completed the first disease response assessment.

After the initiation of trial treatment, safety parameters will be evaluated throughout the study. Adverse event (AE) will be graded according to the National Cancer Institute Common Toxicity Criteria for Adverse Events version 4.0 (NCI CTC AE v4). AE and serious AE (SAE) will be detected and recorded on the Case Report Forms (CRFs) until 15-28 days after the last dose of PEG-BCT-100.

Patients who achieve complete remission (CR)/complete remission with incomplete blood count recovery (CRi) following the 4 consecutive 1600U/kg doses may continue PEG-BCT-100 at the discretion of the investigator.

Patients who achieve partial remission (PR) or stable disease (SD) following the 4 consecutive 1600U/kg doses can continue treatment up to disease progression. Further continuation will be determined by the clinical judgment of the Investigator. Patients who have disease progression will be discontinued PEG-BCT-100.

Blood samples for PK and PD analysis will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 1 to 17 year-old, inclusive.
* Confirmed relapsed/refractory leukemia or lymphoma to the last regimen, and the patient is without standard therapy for the disease.
* For subjects aged <16 years, modified Lansky Play Performance Scale (Appendix A) of 40% or above; For subjects aged ≥16 years, Karnofsky Performance Status (Appendix B) of 40% or above.
* For lymphoma patients, at least one node or nodal mass is measurable by CT scan.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Subject's legally acceptable representative must has signed an informed consent document and patient aged 7 or above must provide an assenting signature on the informed consent document, indicating that he/she/they understand(s) the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

* Has received cancer treatment, e.g. chemotherapy, targeted biologic or enzymes, either approved or investigational, within 2 weeks prior to the start of the PEG-BCT-100.
* Any toxic effects (except hair loss) of the prior therapy have not been resolved to Grade 2 or less according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events.
* Total bilirubin > 1.5 x ULN not related to hemolysis or Gilbert's disease, and AST/ALT > 5 x ULN
* Serum creatinine > 2 x ULN or calculated creatinine clearance < 60 ml/min.
* Any other active malignancy within the past year except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* History of HIV-1 seropositivity.
* Active infection not adequately responding to appropriate therapy.
* Female patient is pregnant or lactating.
* Female patient with childbearing potential and sexual activity who does not agree or unable to use adequate contraceptive [including prescription oral contraceptives (birth control pills), contraceptive injections, intrauterine device (IUD), double-barrier method (spermicidal jelly or foam with condoms or diaphragm), contraceptive patch, or surgical sterilization] before entry and throughout the study.
* Male patient with sexual activity who does not agree to use adequate contraception (barrier method of birth control in conjunction with spermicidal jelly) prior to study entry and throughout the study.
* Use of any investigational drug(s) within 2 weeks prior to the start of the PEG-BCT-100.
* Use of any arginine depleting agent within 2 weeks prior to the start of the PEG-BCT-100.
* Subjects, who in the opinion of the Investigator, are unable to comply with the trial treatment and the related trial procedures.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
safety of PEG-BCT-100 in patients with relapsed or refractory leukemia or lymphoma receiving PEG-BCT-100 | 6 weeks
  The primary endpoint is defined as the adverse event and serious adverse event related to the trial treatment. The adverse event includes unexpected clinical findings which could be related to the metabolic consequences of acute or prolong arginine depletion.
  The following measures will be used to evaluate the safety of the trial treatment:
  1. vital signs
  2. laboratory tests of safety i.e. hematology, blood biochemistry, urinalysis
  3. Adverse events (NCI CTC AE, version 4.0)

SECONDARY OUTCOMES:
efficacy of PEG-BCT-100 in disease control in patients with leukemia or lymphoma who have received 4 doses PEG-BCT-100 1600 U/kg. | 6 days after the first 4 doses of 1600 U/kg PEG-BCT-100
  The percentage of patients who have disease controlled following the 4 doses of PEG-BCT-100 1600 U/kg. Disease control is defined by achieving complete remission (CR) or complete remission with incomplete blood count recovery (CRi) or partial remission (PR), or stable disease (SD).
pharmacokinetics (PK) profiles of PEG-BCT-100. | 1st dose: 1, 72, 168 hrs post dose; 2nd-4th dose: 1, 168 hrs post dose
  The subtracting baseline (SB) method will be used considering the endogenous background of arginase when estimating the PK parameters. The peak and trough concentrations will be listed for each dosing. The elimination rate and half life of rhArg1 will be estimated by the PK samplings during the postponement of trial treatment. The elimination rate will be assumed to be linear and estimated using the non-compartmental model. The individual steady state will be determined by visual inspection.
pharmacodynamics (PD) profiles in terms of plasma arginine in response to PEG-BCT-100. | predose; 1st induction: 1, 2, 4, 71, 168hrs post dose; 2nd induction: 2, 72, 168 hrs post dose; first dose: 1, 72, 168 hrs post dose; 2nd-4th dose: 168hrs post dose
  1. The time to effective plasma arginine depletion defined as plasma arginine < 8uM for the first dose (500 U/kg);
  2. The effectiveness of maintaining effective arginine depletion up to 8 days after multiple doses;
  3. The concentration of plasma arginase during effective arginine depletion.
time to progression in leukemia or lymphoma patients receiving PEG-BCT-100 | 1 year
  measured from date of first dose of PEG-BCT-100 until documention of disease pregression. Death due to cause other than progression will be censored. Patient without an event will be censored at date last known progression-free

CONTACTS AND LOCATIONS:
Overall Officials: Alan K Chiang, Dr., Principal Investigator — Department of Paediatrics and Adolescent Medicine, The University of Hong Kong
Locations (1):
- Department of Paediatrics and Adolescent Medicine, The University of Hong Kong, Hong Kong, China

REFERENCES:
- See also: Clinical Trail Centre, The University of Hong Kong — http://www.hkuctc.com/index.php
- See also: Bio-Cancer Treatment International Limited — http://www.bio-cancer.com/